CLINICAL TRIAL: NCT06460168
Title: Comparative Effects of Mulligan and Maitland Techniques on Pain, Range of Motion and Functional Disability in Post Prp Knee Osteoarthritis
Brief Title: Mulligan and Maitland Techniques in Post PRP Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/01102
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee joint; exercise; Mulligan exercise; Osteoarthritis; prp
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity; Osteoarthritis; Insomnia, Fatal Familial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mulligan(MWM) Technique (Experimental): Group of post prp knee osteoarthritis patients are given Mulligan (MWM) Mobilization technique
  Interventions: Other: Mulligan(MWM) MobilizationTechnique
- Maitland Technique (Active Comparator): Patients are given Maitland Mobilization technique.
  Interventions: Other: Maitland Mobilization technique
- Baseline treatment (No Intervention): This group are given baseline treatment.

INTERVENTIONS:
Other: Mulligan(MWM) MobilizationTechnique — Mulligan Mobilization program in MWM , a therapist-applied pain free accessory gliding force combined with active movement.
  No Of Sessions Per Week: 3 Per Weeks for 6 weeks (50 Min per Session) No of repetitions; 3 sets for 10 repetitions with 1 minute rest between sets.
  Arms: Mulligan(MWM) Technique
Other: Maitland Mobilization technique — will receive (Maitland mobilization program manipulative physiotherapy in which chain of oscillatory joint mobilization grades l-lV based on the pathological limit of tissue are used) In this, the exercises will be performed in 3 sets and 10 repetitions with 5-10s hold and 30s to 1min rest between repetitions.
  No Of Sessions Per Week: 3 Per Weeks for 6 weeks (50 Min per Session)
  Arms: Maitland Technique

SUMMARY:
Knee osteoarthritis (OA) is a major cause of disability nowadays. Osteoarthritis (OA), also known as degenerative joint disease, is typically the result of wear and tear and progressive loss of articular cartilage. It is most common in elderly people and can be divided into two types, primary and secondary. Platelet-rich plasma (PRP) is an autologous blood product that contains a high concentration of platelets, specifically, 3 to 5 times that of normal blood. PRP contains a high concentration of autogenous growth factors, including vascular endothelial growth factor, platelet-derived growth factor, and transforming growth factor-β, which promote the proliferation of chondrocytes and the synthesis of the extracellular matrix. PRP is increasingly being used in the field of sports injury because of its simple preparation method, low cost, and high degree of safety A randomized clinical trial will be conducted at Ibne Sina Hospital,Multan. Non probability convenience sampling technique will be applied to enroll patients who will be allocated through computerized randomization into group A & group B to collect data. Sample size will be 36. This will be allocated to three groups through lottery method. Group A will be given MWM and group B will be given Maitland techniques while Group C will receive only baseline treatment. The study will be completed within the time duration of ten months. Primary Outcome measures of the research will be Pain, Range of motion, functional status. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

DETAILED DESCRIPTION:
A study conducted since 2022 evaluated the comparative effects of muscle energy and mobilization with movement techniques for knee pain, Range of motion and functional disability in patients with knee Osteoarthritis.A randomized clinical trial was conducted at Physiotherapy Department of Bakhtawar Amin College of Rehabilitation Sciences, Multan. Patients of age 40-60 years with active pain for more than 3 months diagnosed with Grade I, II and III of knee osteoarthritis by orthopedic surgeon according to Kellgren and Lawrence Scale and on basis of radiograph were included. Patients with knee osteoarthritis of grade IV, history of fracture dislocation or radiating pain were excluded. Sixty-eight (68) patients were equally divided in two groups Mulligan group and METs group. Pain intensity was 0.19 (p<0.01), WOMAC score was 0.007(p<0.01) Knee flexion was 0.110(P<0.995) and Knee extension deficit score was 0.087 (P<0.998). Coefficient alpha for with in group subject effect for pain, functional disability and knee flexion and extension deficit is (P≤0.05). Both techniques post isometric relaxation technique of METs and mobilization with movement technique of Mulligans significantly reduced pain, functional disability and symptoms .

Since 2022 conducted a study to find out find whether neuromuscular stimulation of vastus medialis oblique (VMO) in combination with Maitland's mobilization and exercises was more effective as compared to Maitland's mobilization with exercises alone in patients with knee OA. Sixty patients with knee OA were purposively selected and randomly distributed to two groups that received an intervention for eight weeks. Group A patients received Maitland's mobilization in combination with exercises and group B patients received the same intervention as group A in combination with neuromuscular stimulation of VMO muscle. Both groups showed significant (P<0.05) within-group improvement in the knee pain levels and stiffness as reflected by NPRS and WOMAC index.

Another study conducted in 2020 investigate the effectiveness of Mulligan's mobilization with movement (MWM) and Myofascial release on pain, range of motion and functional abilities in patients with knee osteoarthritis. A purposive sample of 30 patients from two major hospitals of Faisalabad was randomly divided into two treatment groups. Group A, received Mulligan's MWM and group B received Myofascial release. Electrotherapy and exercise program was the same for both groups. The interventional program was of two weeks (five days a week, once a day). lease were effective for knee osteoarthritis in terms of pain, range of motion, and for functional abilities. However, Mulligan's MWM produced more quick outcomes than Myofascial release.

One study conducted in 2019 study is to determine the outcome and efficacy of Mulligan's mobilization with movement (MWM) with Maitland mobilization along with conventional therapy in the patients with knee osteoarthritis (OA). randomized controlled trial study was performed at the Department of Physiotherapy, Mayo Hospital, Lahore, Pakistan. Sixty-two patients were selected for the study. MWM was introduced in half of the patients and Maitland mobilizations in the second half for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age group 28-55 years
* Male and female
* Grade 2,3,4 of knee osteoarthritis
* Post PRP Osteoarthritic knee joints included
* After 1st month of Post PRP, patients will be included in study

Exclusion Criteria:

* History of surgery of the affected knee
* Infection
* Malignancy
* Non Osteoarthritic joints excluded

Ages: 28 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating scale(NPRS) | 6 weeks
  The Numeric Pain Rating Scale (NPRS) is used to assess pain. On an 11-point Numeric scale, 0 represents the least amount of pain (no pain) and 10 Represents the most amount of pain (worst pain)
Range of motion(ROM) | 6 weeks
  It is frequently employed as a benchmark technique for the assessment of (ROM) as the main component of all joint motions. The range of mobility of a joint is measured using a device known as a goniometer. Goniometry is the art and science of measuring the joint ranges in every plane of the joint. Short arm and long arm versions of the universal goniometer are available. Goniometric measurements are highly reliable provided measurements are conducted by the same therapist. Knee ranges will be taken by a Universal Goniometer
Functional disability | 6 week
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.

CONTACTS AND LOCATIONS:
Overall Officials: Muqaddas Shareef, DPT, Principal Investigator — Riphah International University
Locations (1):
- Ibne Sina Hospital Multan, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burmester GR, Bijlsma JWJ, Cutolo M, McInnes IB. Managing rheumatic and musculoskeletal diseases - past, present and future. Nat Rev Rheumatol. 2017 Jul;13(7):443-448. doi: 10.1038/nrrheum.2017.95. Epub 2017 Jun 15. PMID 28615732
- [Background] Yin P, Jiang Y, Fang X, Wang D, Li Y, Chen M, Deng H, Tang P, Zhang L. Cell-Based Therapies for Degenerative Musculoskeletal Diseases. Adv Sci (Weinh). 2023 Jul;10(21):e2207050. doi: 10.1002/advs.202207050. Epub 2023 May 18. PMID 37199688
- [Background] Shah S, Danda D, Kavadichanda C, Das S, Adarsh MB, Negi VS. Autoimmune and rheumatic musculoskeletal diseases as a consequence of SARS-CoV-2 infection and its treatment. Rheumatol Int. 2020 Oct;40(10):1539-1554. doi: 10.1007/s00296-020-04639-9. Epub 2020 Jul 14. PMID 32666137
- [Background] Bruyere O, Honvo G, Veronese N, Arden NK, Branco J, Curtis EM, Al-Daghri NM, Herrero-Beaumont G, Martel-Pelletier J, Pelletier JP, Rannou F, Rizzoli R, Roth R, Uebelhart D, Cooper C, Reginster JY. An updated algorithm recommendation for the management of knee osteoarthritis from the European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases (ESCEO). Semin Arthritis Rheum. 2019 Dec;49(3):337-350. doi: 10.1016/j.semarthrit.2019.04.008. Epub 2019 Apr 30. PMID 31126594
- [Background] Diez-Perez A, Brandi ML, Al-Daghri N, Branco JC, Bruyere O, Cavalli L, Cooper C, Cortet B, Dawson-Hughes B, Dimai HP, Gonnelli S, Hadji P, Halbout P, Kaufman JM, Kurth A, Locquet M, Maggi S, Matijevic R, Reginster JY, Rizzoli R, Thierry T. Radiofrequency echographic multi-spectrometry for the in-vivo assessment of bone strength: state of the art-outcomes of an expert consensus meeting organized by the European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases (ESCEO). Aging Clin Exp Res. 2019 Oct;31(10):1375-1389. doi: 10.1007/s40520-019-01294-4. Epub 2019 Aug 17. PMID 31422565
- [Background] O'Connell NE, Smith KJ, Peterson MD, Ryan N, Liverani S, Anokye N, Victor C, Ryan JM. Incidence of osteoarthritis, osteoporosis and inflammatory musculoskeletal diseases in adults with cerebral palsy: A population-based cohort study. Bone. 2019 Aug;125:30-35. doi: 10.1016/j.bone.2019.05.007. Epub 2019 May 8. PMID 31075418
- [Background] Bonanni R, Cariati I, Tancredi V, Iundusi R, Gasbarra E, Tarantino U. Chronic Pain in Musculoskeletal Diseases: Do You Know Your Enemy? J Clin Med. 2022 May 6;11(9):2609. doi: 10.3390/jcm11092609. PMID 35566735